CLINICAL TRIAL: NCT06531174
Title: Exploring Individual Nutrition Care Elements and Nutritional Evaluation Methods Within Dietetic Practice in Cancer Care
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 240901
Record Dates: First submitted 2024-07-22; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cancer; Malnutrition
MeSH Terms: conditions — Neoplasms; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to explore and deepen the understanding of the dietitian's role and work related to individually tailored nutritional treatment in cancer care. The research questions focus on behavior change strategies, goal setting, the possibility of using calf circumference to assess changes in muscle mass, and mapping energy and protein intake, nutritional symptoms, and food-related quality of life during nutritional treatment for cancer patients.

In the first part of the project, audio recordings of conversations between dietitians and patients with cancer will be conducted to investigate the dietitian's work with behavior change strategies and goal setting. Data analysis will be performed using two different methods: content analysis and thematic analysis. The research subjects include both dietitians and cancer patients who engage in conversations.

The second part of the project will include 100 patients with cancer at risk for or with malnutrition. Data collection will involve measurements of weight, height, calf circumference, muscle mass, energy and protein intake, nutritional symptoms, and food-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the first part of the project involve encountering dietitians treating patients with cancer who have malnutrition or are at risk of malnutrition. For these patients, the inclusion criteria are as follows:

* aged ≥18 years with a diagnosed cancer
* ongoing nutrition therapy by a dietitian
* malnutrition or risk of malnutrition according to the hospitals criteria where at least one of the following criteria must be met: low BMI, involuntary weight loss, and/or eating difficulties. Patients can also be included if they are referred to a dietitian based on treatment guidelines due to a high risk of malnutrition associated with the cancer diagnosis or its medical therapy.

For the second part of the project, the inclusion criteria are:

* aged ≥18 years with a diagnosed cancer
* undergoing or planned treatment, including surgical, oncological, or a combination of these
* have been referred to a dietitian but have not yet had their initial contact with the dietitian, and
* malnutrition or risk of malnutrition according to the hospital's criteria, where at least one of the following criteria must be met: low BMI, involuntary weight loss, and/or eating difficulties. Patients can also be included if they are referred to a dietitian based on treatment guidelines due to a high risk of malnutrition associated with the cancer diagnosis or its medical therapy.

Exclusion Criteria:

For the first part of the project, the exclusion criteria regarding patients are:

* known dementia or impaired cognitive function, and
* not proficient in spoken and written Swedish.

For the second part of the project, the exclusion criteria are:

* known dementia or impaired cognitive function,
* ongoing nutrition therapy by a dietitian at inclusion, and
* not proficient in spoken and written Swedish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the first part of the project (non-probability sampling method), research participants are registrered dietitians in Sweden and patients with cancer who have malnutrition or are at risk of malnutrition. The participants are recruited systematically through a strategic or purposive selection within the hospital setting.
  For the second part of the project (probability sampling method), research participants are patients aged ≥18 years with a diagnosed cancer who are receiving or scheduled to receive treatment, including surgical, oncological, or a combination of these, at Uppsala University Hospital in Uppsala. The patients should have been referred to a dietitian but have not yet had their initial contact with the dietitian at the time of inclusion.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Calf Circumference | Baseline, 1 month and 3 months
  Measured on right and left calf

SECONDARY OUTCOMES:
Fat Free Mass and Fat Mass | Baseline, 1 month and 3 months
  Measured with bioimpedance analysis
Food-Related Quality of Life | Baseline, 1 month and 3 months
  Measured with the questionnaire Satisfaction with Food-Related Life. This instrument contains seven statements where the participant responds on a seven-point scale from 'Strongly disagree' to 'Strongly agree'. A higher rating indicates a worse outcome.
Energy and Protein Intake | Baseline, 1 month and 3 months
  Measure with a repeated 24 h recall interview
Nutrition Impact Symptoms | Baseline, 1 month and 3 months
  Measured with the Eating Symptoms Questionnaire (13 symtoms to be rated on a five-level scale from no trouble at all to severe) and the Disease-Related Appetite Questionnaire (11 questions about appetite, hunger and other symtoms). A higher number of symtoms indicates a worse outcome.
Quality of Life | Baseline, 1 month and 3 months
  Measured with the instrument EORTC QLQ-C30. Includes 28 symptoms or issues, each rated on a four-level scale from 1= 'not at all' to 4 = 'very much. A higher score indicates a worse outcome. The lowest aggregated score of the instrument is 28 and the highest is 112. The instrument also contains two questions where one is to rate their overall health and quality of life on a seven-level scale from 1= 'Very poor" to 7= 'Excellent'.
Muscle Function and Strength | Baseline, 1 month and 3 months
  Measured with 30s chair stand test and hand dynamometer

OTHER OUTCOMES:
Categories and frequencies of Behaviour Change Strategies | Baseline
  For part 1 of the project, data is collected by conversation recordings. The behaviour change taxonomy (v1) by Miche et al (2013) will be used to categorize and count the strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Evelina Liljeberg, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No